CLINICAL TRIAL: NCT07094334
Title: Investigation of the Acute Effects of a Single Session of Action Observation and Motor Imagery Training on Upper Extremity Balance, Muscle Oxygenation, and Fatigue in Young Adults
Brief Title: Investigation of Single Session Action Observation and Motor Imagery Training on Balance, Muscle Oxygenation, Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Eren Ozen, Principal Investigator, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025 - 904
Record Dates: First submitted 2025-07-19; First posted 2025-07-30 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Motor Imagery Training; Action Observation Training
Keywords: Motor imagery training; Action observation training; muscle oxygenation; fatigue; upper extremity balance; acute effect
MeSH Terms: conditions — Fatigue | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Action Observation Group (Experimental): Prior to the intervention, the Upper Extremity Closed Kinetic Chain Stability Test will be administered to determine participants' upper extremity balance levels. Participants in the group will watch video recordings of the Upper Extremity Closed Kinetic Chain Stability Test, performed by a third person, from various angles, at both normal and slow motion speeds, for a total duration of 10 minutes. Following the intervention, the Upper Extremity Closed Kinetic Chain Stability Test will be performed in four repetitions, identical to the pre-intervention assessment. In order to prevent fatigue from influencing the outcomes, participants will be given a 5-minute rest period between the pre- and post-intervention assessments. The Moxy device will continuously monitor throughout all procedures. The fatigue levels of the participants will be evaluated prior to and following the test.
  Interventions: Other: Action Observation
- Action Observation combined with Motor Imagery Group (Experimental): Prior to the intervention, the Upper Extremity Closed Kinetic Chain Stability Test will be administered to determine participants' upper extremity balance levels. Participants in this group will be asked to imagine themselves performing the Upper Extremity Closed Kinetic Chain Stability Test while watching video recordings of the test, captured from different angles and executed by a third person, for a total duration of 10 minutes at both normal and slow-motion speeds. Following the intervention, the Upper Extremity Closed Kinetic Chain Stability Test will be performed in four repetitions, identical to the pre-intervention assessment. In order to prevent fatigue from influencing the outcomes, participants will be given a 5-minute rest period between the pre- and post-intervention assessments. The Moxy device will continuously monitor throughout all procedures. The fatigue levels of the participants will be evaluated prior to and following the test.
  Interventions: Other: Action Observation combined with Motor Imagery
- Control Group (Sham Comparator): Prior to the intervention, the Upper Extremity Closed Kinetic Chain Stability Test will be administered to determine participants' upper extremity balance levels. The participants will watch landscape and nature-themed videos for a duration of 10 minutes. Following the intervention, the Upper Extremity Closed Kinetic Chain Stability Test will be performed in four repetitions, identical to the pre-intervention assessment. In order to prevent fatigue from influencing the outcomes, participants will be given a 5-minute rest period between the pre- and post-intervention assessments. The Moxy device will continuously monitor throughout all procedures. The fatigue levels of the participants will be evaluated prior to and following the test.
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Other: Action Observation — This study, in contrast to prior research, will examine both the acute effects of action observation therapy and its impacts at the peripheral level.
  Arms: Action Observation Group
Other: Action Observation combined with Motor Imagery — This study, in contrast to prior research, will examine both the acute effects of action observation therapy combined with motor imagery and its impacts at the peripheral level.
  Arms: Action Observation combined with Motor Imagery Group
Other: Sham (No Treatment) — Participants in this intervention group will watch landscape and nature-themed videos for the duration corresponding to the intervention period applied in the other groups.
  Arms: Control Group

SUMMARY:
Action observation (AO) and motor imagery (MI) interventions are frequently employed both in the rehabilitation process following orthopedic injuries and surgeries, with aims such as reducing pain and increasing joint range of motion, as well as in the rehabilitation of neurological disorders to restore motor functions and achieve functional independence. In recent years, it has been demonstrated that AO and MI training can exert positive effects on motor performance and neurophysiological activation. Notably, when AO and MI training are applied in combination, it has been suggested that they produce a more pronounced impact on motor performance and support motor learning processes. The effects of these techniques have generally been evaluated following long-term interventions, and there is limited data in the literature regarding their effects after a single session. Furthermore, it has been shown in the literature that action observation and motor imagery training can elicit cortical activation. However, current scientific evidence concerning the peripheral effects of these interventions remains limited. Therefore, the aim of the present study is to investigate the acute effects of a single session of action observation and motor imagery training on upper extremity balance, muscle oxygenation, and fatigue in asymptomatic young adult males

ELIGIBILITY:
Inclusion Criteria:

* To be between 18 and 25 years of age
* To have no history of any surgical procedure involving the upper extremity
* To be male**

  * Since the Upper Extremity Closed Kinetic Chain Stability Test is conducted in a different position for females, only male participants will be included in the study to maintain group homogeneity.

Exclusion Criteria:

* Scoring 24 or below on the Mini Mental State Examination (MMSE)
* Having hearing, visual, or perceptual impairments that may affect the study outcomes
* Presence of any upper extremity problem
* Having neurological, metabolic, or systemic diseases

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Closed Kinetic Chain Stability Test | Before Intervention
  In this test, participants assume a push-up position, positioned between two parallel strips placed on the floor, and touch the opposite strips in a cross-body manner with their hands for 15 seconds. The total number of touches is recorded as the score. The test is performed four times, with a 45-second rest interval between each trial. The participant's test score is calculated as the average of the scores from the last three trials.
Upper Extremity Closed Kinetic Chain Stability Test | immediately after the intervention
  In this test, participants assume a push-up position, positioned between two parallel strips placed on the floor, and touch the opposite strips in a cross-body manner with their hands for 15 seconds. The total number of touches is recorded as the score. The test is performed four times, with a 45-second rest interval between each trial. The participant's test score is calculated as the average of the scores from the last three trials.

SECONDARY OUTCOMES:
Muscle oxygenation | Before Intervention
  In this study, the Moxy Monitor device will be used to assess the upper extremity muscle oxygenation levels of the participants. This device operates using near-infrared spectroscopy (NIRS) technology and non-invasively measures the amounts of oxygenated and deoxygenated hemoglobin in muscle tissue. The validity and reliability of the Moxy Monitor device in physiological measurements have been reported in numerous studies. Measurements will be conducted by placing the sensor on the anterior portion of the deltoid muscle on the participants' dominant side.
Muscle Oxygenation | immediately after the intervention
  In this study, the Moxy Monitor device will be used to assess the upper extremity muscle oxygenation levels of the participants. This device operates using near-infrared spectroscopy (NIRS) technology and non-invasively measures the amounts of oxygenated and deoxygenated hemoglobin in muscle tissue. The validity and reliability of the Moxy Monitor device in physiological measurements have been reported in numerous studies. Measurements will be conducted by placing the sensor on the anterior portion of the deltoid muscle on the participants' dominant side.
Modified Borg Scale | pre-intervention
  Participants will rate their level of fatigue on a scale ranging from 0 (no fatigue at all) to 10 (maximum fatigue).
Modified Borg Scale | immediately after the intervention
  Participants will rate their level of fatigue on a scale ranging from 0 (no fatigue at all) to 10 (maximum fatigue).

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Hazar, Prof., Study Director — Gazi University; Sıla Çağla Demiralay, M.Sc., Study Chair — Gazi University; Şeyma CEBE KARACA, M.Sc., Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)